CLINICAL TRIAL: NCT01136044
Title: Clinical Experience With a Tensor Fasciae Latae Perforator Flap Based on Septocutaneous Perforators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Dr.Martin Hubmer, Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUG111
Record Dates: First submitted 2010-05-28; First posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Soft Tissue Defect
Keywords: tensor fasciae latae; septocutaneous perforators
MeSH Terms: interventions — Perforator Flap

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: septocutaneous perforator flap — Perforator flaps can be based on septocutaneous or musculocutaneous perforators. If septocutaneous perforators are present, the harvest of these flaps is more straight forward and the dissection of the pedicle is easy.
  Other Names: fasciocutaneous flaps; perforator flap

SUMMARY:
The purpose of this study is to evaluate the possible harvest of a tensor fasciae latae flap based on septocutaneous perforators.This study should further confirm our data from an anatomical study concerning location, distribution, diameter and differentiation of the perforators.

ELIGIBILITY:
Inclusion Criteria:

* soft tissue defect
* no previous operations in the thigh region

Exclusion Criteria:

* obese patients

Ages: 16 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Confirmation of the anatomical data in the clinical trial | January 2008 till may 2010
  Since the purpose of this study was to confirm our anatomical data in a clinical trial, the location, the differentiation and the diameter of the septocutaneous perforators has been measured and recorded during flap elevation.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hubmer, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Surgery, Division of Plastic Surgery, Graz, Austria

REFERENCES:
- [Background] Hubmer MG, Schwaiger N, Windisch G, Feigl G, Koch H, Haas FM, Justich I, Scharnagl E. The vascular anatomy of the tensor fasciae latae perforator flap. Plast Reconstr Surg. 2009 Jul;124(1):181-189. doi: 10.1097/PRS.0b013e3181ab114c. PMID 19568071